CLINICAL TRIAL: NCT07084194
Title: Impact of Integrating Two Nano Based Irrigants With Two Activation Techniques in Treatment of Teeth With Acute Pulpitis on Postoperative Pain and Flare up Incidence: A Randomized Clinical Study
Brief Title: Impact of Integrating Two Nano Based Irrigants With Two Activation Techniques in Treatment of Teeth With Acute Pulpitis on Postoperative Pain and Flare up Incidence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Rabee Ibrahaim Ismail Alhabibi, Rabee Alhabibi, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EC Reaseach NO.1079
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Flare up; Flare Up, Symptom
Keywords: postoperative pain; flare up; nano-technology; irrigation; chitosan; aloe-vera
MeSH Terms: conditions — Pain, Postoperative; Symptom Flare Up

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP I (Experimental): treated with nanochitosan and passive ultrasonic activation
  Interventions: Other: Chitosan Nanoparticles Irrigant; Device: ultrasonic activator
- GROUP II (Experimental): treated with nanochitosan and laser activation
  Interventions: Other: Chitosan Nanoparticles Irrigant; Device: Diode Laser Activation
- GROUP III (Experimental): treated with nano-Aloe Vera and passive ultrasonic activation
  Interventions: Other: aloe vera nanoparticles irrigant; Device: ultrasonic activator
- GROUP IV (Experimental): treated with nano-Aloe Vera and laser activation
  Interventions: Other: aloe vera nanoparticles irrigant; Device: Diode Laser Activation

INTERVENTIONS:
Other: Chitosan Nanoparticles Irrigant — using Chitosan Nanoparticles irrigant as a final irrigation solution.
  Arms: GROUP I; GROUP II
Other: aloe vera nanoparticles irrigant — using Aloe Vera Nanoparticles irrigant as a final irrigation solution.
  Arms: GROUP III; GROUP IV
Device: Diode Laser Activation — activation of nanoparticles irrigants using diode laser
  Arms: GROUP II; GROUP IV
Device: ultrasonic activator — activation of nanoparticles irrigants using ultrasonic activator
  Arms: GROUP I; GROUP III

SUMMARY:
This study aimed to evaluate and compare impact of integrating passive ultrasonic activation and laser activation with nano-chitosan and aloe vera in terms of postoperative pain and flare-up incidence in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 (adults only)
* multiple-rooted with multiple root canal.
* Permanent teeth with mature apex and complete root formation.
* Without root caries.
* Tooth must be restorable.
* Without anatomical abnormalities such as fusion.
* Healthy patient category I according to ASA.
* Vital tooth, with acute irreversible pulpitis and without peri-apical periodontitis.
* No periapical radiolucency.
* Consent Patients for who consent to participate and attend follow-up appointments.

Exclusion Criteria:

* single root canals or double root.
* Root canal calcifications.
* Root resorption or fracture.
* Previously root canal treated teeth.
* immunocompromised patients.
* Pregnant females
* Patients with systemic diseases as diabetic or hypertension patients.
* Patients with facial swelling.
* patients who use analgesics or antibiotics within 48-72 hours.
* Allergy to any materials used (e.g., irrigants or anesthetics).
* psychiatric illness
* Teeth that are not indicated for endodontic treatment: bad oral hygiene, mobile teeth, or recessed teeth.
* Previously endodontically treated teeth.
* Teeth with sinus tract.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
postoperative pain intensity Postoperative pain is to be assessed using visual analog scale (VAS), A scale from (0 to 10) where "0" means no pain and "10 means a severe pain that has never faced before. | [Time Frame: 6, 12, 24, 48, 72 hours and 7 days after the first visit to collect the postoperative pain data.]
  Patients will be contacted by phone at 6, 12, 24, 48, 72 hours and 7 days after the first visit to collect the postoperative pain data.

SECONDARY OUTCOMES:
Flare-Up Incidence Flare-up is assessed through asking the patient to notify the investigator if any sudden severe pain or swelling takes place. | [Time Frame: Within 7 days post-treatment)
  This could require an unscheduled emergency visit or prescription of additional medication.

IPD SHARING:
Plan to Share IPD: Undecided